CLINICAL TRIAL: NCT05014230
Title: Acute Pain Treatment: A Randomized Controlled Trial Examining Opioids and Open Placebo
Brief Title: Open Label Placebo to Reduce Prescription Opioid Use
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brown University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); The Miriam Hospital (Other); Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2106003017; K01DA048087 (NIH)
Record Dates: First submitted 2021-08-13; First posted 2021-08-20 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Acute Pain
Keywords: pain; placebo; analgesia; opioid
MeSH Terms: conditions — Acute Pain; Pain; Agnosia

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (Other): Opioid medication, as prescribed in routine care
  Interventions: Other: Opioid medication as part of standard care
- Open Label Placebo + Treatment as Usual (Experimental): Opioid medication, as prescribed in routine care + Honest placebos
  Interventions: Dietary Supplement: Open Placebo; Other: Opioid medication as part of standard care

INTERVENTIONS:
Dietary Supplement: Open Placebo — Zeebo
  Arms: Open Label Placebo + Treatment as Usual
Other: Opioid medication as part of standard care — Opioid medication as prescribed by prescriber. This is not impacted by being in the research study.

SUMMARY:
The goal of the proposed study is to examine the efficacy of using an honest placebo to relieve pain for patients with an acute pain condition. People with acute pain will receive their standard dose of opioid medication for pain management. In addition, some people will be asked to take placebo pills, honestly described as placebos, as well. Patients will answer a few short questions over the phone once per day for seven days about pain and opioid use. The investigators hypothesize that participants in the open label placebo group will take fewer opioids and have less pain than those in the treatment as usual group.

DETAILED DESCRIPTION:
America is in the midst of an opioid epidemic. One of the reasons opioid addiction and overdose deaths have recently increased is that doctors are frequently prescribing opioid medication as a treatment for pain. If researchers can develop ways of increasing the pain-relief patients experience from a set amount of opioids, then doctors might ultimately be able to prescribe fewer opioid medications, which could help curb the opioid crisis.

Although "placebos," a medication whose benefit derives solely from positive psychological factors rather than pharmacological factors, are often disparaged in medicine, research suggests that placebos can actually help reduce pain. In fact, there is reason to think that placebos are effective even when a patient knows they are taking a placebo.

The goal of the proposed study is to examine the efficacy of using an honest placebo to relieve pain for patients with an acute pain condition. People with acute pain in the Emergency Department, or patients undergoing hand/wrist surgery, will receive their standard dose of opioid medication for pain management. In addition, some people will be asked to take placebo pills, honestly described as placebos, as well. Patients will answer a few short questions over the phone once per day for seven days regarding their pain, opioid use, and placebo use (only those assigned to take placebo pills).

ELIGIBILITY:
Inclusion

* 18 years or older
* English Speaking
* Has a working smart-phone
* Able to provide informed consent
* Present for upper or lower extremity fracture (ED sample only) or for hand or wrist surgery (hand surgery sample only)
* Are expected to be prescribed opioids at discharge
* Are expected to be discharged from the Emergency Department (ED sample only)
* Intends to take 1 or more doses of opioid medication as prescribed

Exclusion

* Chronic opioid use
* Unlikely to follow-up (discretion of investigator and treating provider)
* Having been diagnosed with a psychotic disorder
* Having a current medical marijuana prescription
* Currently receiving worker's compensation or intending to apply for worker's compensation
* History of opioid use disorder
* Allergy to opioid medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2021-12-09 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Prescription Opioid Use | 7 days
  Quantity of Opioid Use (converted to MME when possible)

SECONDARY OUTCOMES:
Pain Intensity | 7 days
  Pain Intensity subscale of the Brief Pain Inventory
Pain Interference | 7 days
  Pain interference subscale of the Brief Pain Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Bernstein, PhD, Principal Investigator — Brown University
Locations (1):
- Lifespan Hospital System, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No